CLINICAL TRIAL: NCT04781894
Title: Application of Transthoracic Shear-wave Ultrasound Elastography in Pleural Lesions
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202012200RINA
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Elasticity Imaging Techniques
Keywords: Shear wave ultrasound elastography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to provide the information of tissue elasticity in different etiologies of pleural lesions and to validate the predictive value of shear-wave elastography in differentiating benign pleural lesions from malignant lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiographic evidence of pleural lesions or effusion

Exclusion Criteria:

* Age < 20 y/o
* Patients who cannot hold their breath for 5 seconds

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving chest ultrasonography in National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2025-01-25 (Estimated); Study Completion 2025-01-25 (Estimated)

PRIMARY OUTCOMES:
Application of transthoracic shear-wave ultrasound elastography in pleural lesions | six months
  to provide the information of tissue elasticity in different etiologies of pleural lesions and to validate the predictive value of shear-wave elastography in differentiating benign pleural lesions from malignant lesions

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Wen Kuo, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan